CLINICAL TRIAL: NCT01886482
Title: Effect of High Protein Diet on Cardiovascular Diseases Risk Factors Among Overweight and Obese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Isfahan University of Medical Sciences, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: high protein diet in childhood
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Body Mass Index Quantitative Trait Locus 7 Disorder; Tangier Disease
MeSH Terms: conditions — Tangier Disease | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nutrition intervention (Active Comparator): high protein diet
  Interventions: Other: nutrition intervention
- no intervention (No Intervention): control diet

INTERVENTIONS:
Other: nutrition intervention — high protein diet
  Arms: nutrition intervention

SUMMARY:
The investigators aimed to determine the effects of HP diet on CVD risk factors among overweight and obese children.

DETAILED DESCRIPTION:
Background: Studies regarding the effects of high protein (HP) diet on cardiovascular (CVD) risk factors have reported contradictory results.

Objective: In present study, the investigators aimed to determine the effects of HP diet on CVD risk factors among overweight and obese children.

Design: In this randomized controlled trial, the investigators recruited 50 overweight and obese women, aged 6-11years into HP or control energy restricted diets for 10 weeks (protein, carbohydrate, fat: 25%, 45%, 30% vs. 15%, 55%, 30%, respectively). Total protein amount, divided to animal and plant sources in 50%-50% and animal sources distributed (half/half) between meats and dairy products. Fasting blood samples, lipid profile, systolic and diastolic blood pressure and anthropometric measurements were measured based on the standard guidelines.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 85th age of 6-11 years
* no history of chronic diseases
* no taken medications

Exclusion Criteria:

* do not prescribe their diet
* mental retardation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
the amount of weight reduction in two dietary groups | 10 weeks
  weight reduction (kg)

SECONDARY OUTCOMES:
LDL (mg/ml) | 10 weeks
HDL (mg/ml) | 10 weeks
fasting blood glucose | 10 weeks
total cholesterol (mg/dl) | 10 weeks
blood pressure | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran